CLINICAL TRIAL: NCT01667276
Title: Acceptability of Depo-subQ in Uniject
Status: Completed | Type: Observational
Sponsor: FHI 360 (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); PATH (Other)
Responsible Party: Sponsor
Other Study IDs: 10196
Record Dates: First submitted 2012-08-02; First posted 2012-08-17 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Contraception
Keywords: AE adverse event; AIDS acquired immunodeficiency syndrome; ALT (SGPT) alanine aminotransferase; ART antiretroviral therapy; AST (SGOT) aspartate aminotransferase; DCF data collection forms; DMC Data Monitoring Committee; FDA (U.S.) Food and Drug Administration; GCP Good Clinical Practice guidelines; HB sAg Hepatitis B surface antigen; ICH International Conference of Harmonisation; IND Investigational New Drug Application; IRB Institutional Review Board; IU international units; mg milligram(s); mm3 cubic millimeter(s); PCR polymerase chain reaction; SAE serious adverse event; µg microgram; ULN upper limit of the normal range; WB Western Blot
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational study to assess the experience of current depot medroxyprogesterone acetate (DMPA) intramuscular (IM) clients and providers when they try Depo-subQ in Uniject and offer recommendations for the introduction of this method.

DETAILED DESCRIPTION:
This is an observational study to assess the experience of current depot medroxyprogesterone acetate (DMPA) intramuscular (IM) clients and providers when they try Depo-subQ in Uniject and offer recommendations for the introduction of this method.

A total of 560 participants will be enrolled in the study in the following groups:

360 participants (120 in Uganda and 240 in Senegal) who are current DMPA IM clients who seek re-injection of DMPA from either community health workers (CHWs) or clinic-based providers; and are 18-40 years of age; received their most recent DMPA injection no more than 13 weeks prior to enrollment in the study [16].

Up to 100 participants (50 in Uganda and 50 in Senegal) current DMPA IM clients who meet the inclusion/exclusion criteria but do not want to receive the injection with Depo-subQ in Uniject and are willing to complete a short questionnaire

80 CHWs (40 in Uganda and 40 in Senegal) and 20 clinic-based providers (from Senegal only) who are trained to give Depo-subQ in Uniject as part of this study

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40
* In general good health (the participant verbally reports she feels well)
* Using DMPA continuously for at least six months prior to enrollment in the study (i.e., had at least two previous injections)
* Received their most recent DMPA injection no more than 13 weeks prior to enrollment in the study at the study clinic or from a family planning provider involved in the study (Senegal only)
* Received their most recent DMPA injection no more than 13 weeks prior to enrollment in the study from a family planning provider involved in the study (Uganda only)
* Desires to be re-injected with DMPA
* Willing to sign an informed consent document
* Willing to provide contact information and be interviewed three months after enrollment.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 560 participants will be enrolled in the study in the following groups:
  * 360 participants (120 in Uganda and 240 in Senegal) who are current DMPA IM clients who seek re-injection of DMPA from either CHWs or clinic-based providers; and are 18-40 years of age; received their most recent DMPA injection no more than 13 weeks prior to enrollment in the study [16].
  * Up to 100 participants (50 in Uganda and 50 in Senegal) current DMPA IM clients who meet the inclusion/exclusion criteria but do not want to receive the injection with Depo-subQ in Uniject and are willing to complete a short questionnaire
  * 80 CHWs (40 in Uganda and 40 in Senegal) and 20 clinic-based providers (from Senegal only) who are trained to give Depo-subQ in Uniject as part of this study
Sampling Method: Non-Probability Sample
Enrollment: 476 (Actual)
Dates: Start 2012-07; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Measure the acceptability of Depo-subQ in Uniject among DMPA IM family planning clients; | 1 year
  percent of participants who declare they would select Depo-subQ in Uniject for their next injection if this drug product was available at three months with a 95% confidence interval per country
2) Measure the acceptability of Depo-subQ in Uniject among family planning providers (both clinic-based and CHWs); | 1 year
  key themes will be identified from interview transcripts to summarize family planning providers' (clinic-based and CHWs) acceptability of Depo-subQ in Uniject and preference for administering Depo-subQ in Uniject relative to the typical DMPA intramuscular injection by county
Assess family planning providers' (clinic-based and CHWs) training materials. | 1 year
  descriptive analyses (e.g., frequencies and means) of responses for quantitative questions and summaries providers' qualitative responses to open-ended questions from the post-training evaluation for each country

SECONDARY OUTCOMES:
1) To qualitatively compare acceptability of Depo-subQ in Uniject among the two types of family planning providers-clinic-based and CHWs (Senegal only) | 1 year
  frequencies and summary statistics of acceptability data among family planning clients by asking participants to compare their experiences receiving Depo-subQ in Uniject to their experiences receiving the typical DMPA intramuscular injection by country
2) To assess the safety of participants who receive Depo-subQ in Uniject during the study | 1 year
  frequencies of reported adverse events by country

CONTACTS AND LOCATIONS:
Overall Officials: Holly Burke, PhD, MPH, Principal Investigator — FHI 360; Anthony Mbonye, MD, PhD, Principal Investigator — Ministry of Health, Uganda; Bpcar M Daff, MD, PhD, MSc, Principal Investigator — Division de la Sante de la Reproduction
Locations (2):
- Ministry of Health Clinics, All Cities Where There Is A Clinic, Senegal
- Ministry of Health Clinics, Uganda, All Cities Where There Is A Clinic, Uganda

REFERENCES:
- [Derived] Burke HM, Mueller MP, Perry B, Packer C, Bufumbo L, Mbengue D, Mall I, Daff BM, Mbonye AK. Observational study of the acceptability of Sayana(R) Press among intramuscular DMPA users in Uganda and Senegal. Contraception. 2014 May;89(5):361-7. doi: 10.1016/j.contraception.2014.01.022. Epub 2014 Feb 6. PMID 24631328
- [Derived] Burke HM, Mueller MP, Packer C, Perry B, Bufumbo L, Mbengue D, Daff BM, Mbonye A. Provider acceptability of Sayana(R) Press: results from community health workers and clinic-based providers in Uganda and Senegal. Contraception. 2014 May;89(5):368-73. doi: 10.1016/j.contraception.2014.01.009. Epub 2014 Jan 21. PMID 24576792